CLINICAL TRIAL: NCT05562479
Title: Effect of Sars-cov-2 on Donor Oocyte Quality and Quantity, a Multicenter Retrospective Study.
Status: Completed | Type: Observational
Sponsor: Novafem (Other)
Responsible Party: Principal Investigator, Jose Pablo Saffon, Director, Novafem
Other Study IDs: Novafem
Record Dates: First submitted 2022-09-28; First posted 2022-09-30 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Ovarian Reserve; SARS-CoV-2 Infection; Blastocyst
Keywords: COVID-19; SARS-CoV-2; embryos;; endometrium;; female reproductive system; in vitro fertilization;; menstrual cycle;; oocytes;; ovarian reserve; blastocyst
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Non exposed to Sars Cov 2 egg donors: Evaluate the results within oocyte retrieval, oocyte fertilisation and blastocyst formation.
  Interventions: Biological: Sars Cov 2 infection; Biological: Sars Cov 2 vaccination
- Exposed to Sars Cov 2 Infection: Evaluate the results within oocyte retrieval, oocyte fertilisation and blastocyst formation, after being exposed to the infection.
- Exposed to Sars Cov 2 Vaccines: Evaluate the results within oocyte retrieval, oocyte fertilisation and blastocyst formation, after being exposed to vaccination.

INTERVENTIONS:
Biological: Sars Cov 2 infection — Donors recovered from Sars Cov 2 Infection
  Groups: Non exposed to Sars Cov 2 egg donors
Biological: Sars Cov 2 vaccination — Egg Donors vaccinated
  Groups: Non exposed to Sars Cov 2 egg donors

SUMMARY:
Purpose: To determine the impact of SARS-CoV-2 infection and immunization on ovarian response to controlled ovarian stimulation (COS) and embryo development after in vitro fertilization (IVF) Methods: A retrospective multicentric cohort study of 427 oocyte donors was conducted between January 1st, 2018 and September 18th, 2022. Patients who recovered from SARS-CoV-2 infection, vaccinated or non-exposed were included. Demographic, cycle characteristics, and laboratory outcomes were compared.

DETAILED DESCRIPTION:
This was a multicenter retrospective cohort study performed at the Centro de Fertilidad y Genetica Novafem, Bogota, Colombia, and Clinica de la Mujer - Medicina Reproductiva, Viña del Mar, Chile. The Ethics Committee approved the study protocol of both centers. Informed contents were obtained from patients for data collection with scientific use.

All donors who underwent COS for oocyte donation between January 1st, 2018 and July 31th, 2022 were screened for eligibility and followed up to September 18th, 2022.

Oocyte donation cycles were utilized because this model is an excellent choice for controlling known female characteristics. Previous research concluded that a major predictor of ART outcomes is maternal age.

Eligibility criteria were donors aged older than 18 years or younger than 35 years. After providing informed consent, the patients were questioned about their confirmed past SARS-Cov-2 infection/vaccination status. Patients were categorized into the vaccinated group if they had received two dosages of any SARS-CoV-2 vaccines (BNT162b2 mRNA Pfizer-Biontech, mRNA-1273 Moderna or inactivated SARS-CoV-2 vaccine Sinovac) with a break of at least three weeks between each dose. First and second vaccine dates were requested of vaccinated patients. Vaccine administration details, such as vaccine type, dose, date, manufacturer, and lot number, were collected from immunization records.

For recovering patients, the date of a negative nasopharyngeal COVID polymerase chain reaction (PCR) test was registered. None of the recovering patients were vaccinated with any SARS-CoV-2 vaccine. Both clinics strictly required a negative PCR test for SARS-CoV-2 RNA detection 5 days before oocyte retrieval, except for those patients who were less than 3 months following recovery from SARS-Cov-2 infection. Patients in the control group were selected from medical records prior to March 2020 to ensure they did not have the infection and were not vaccinated.

Data including the patient age, body mass index (BMI), antral follicle count (AFC), anti mullerian hormone (AMH), days of stimulation, average dose of gonadotropins, the number of retrieved oocytes, mature oocytes, fertilized oocytes and top quality embryos obtained were recorded. Other parameters were calculated such as the ratio between the number of retrieved oocytes and the number of mature follicles in order to assess the adequacy of response of the follicle to the LH/hCG trigger; the fertilization rate (FR), which was defined as the proportion of inseminated oocytes with 2PN at the time of the fertilization check on Day 1 and finally the blastocyst development rate, defined as the proportion of 2PN zygotes which are at the blastocyst stage at Day 5.

All analyses were performed using SPSS 23.0 (SPSS Inc., Chicago, IL, USA). Normally, distributed data were compared across study groups by univariate ANOVA. All P-values were tested as two-tailed and considered significant at <0.05.

ELIGIBILITY:
Inclusion

* Age: 18 - 32 Years
* Body Mass Index between 18 and 26
* AFC: Antral follicular count over 15 in total.
* AMH: Anti-Mullerian hormone over 2.5
* Signed consents.
* Covid vaccines and infection information (for case group).

Exclusion:

* Egg donors with incomplete information of days of stimulation, average dose of gonadotropins, the number of retrieved oocytes, mature oocytes, fertilised oocytes and top-quality embryos obtained.
* Familial genetic disorders.
* Menstrual cycle disorders.
* Polycystic ovary syndrome.

Ages: 18 Years to 32 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients were categorized into the vaccinated group if they had received two dosages of any SARS-CoV-2 vaccines with a break of at least three weeks between each dose. First and second vaccine dates were requested from vaccinated patients. Vaccine administration details, such as vaccine type, dose, date, manufacturer, and lot number, were collected from immunization records.
  For recovering patients, the date of an adverse nasopharyngeal COVID polymerase chain reaction (PCR) test was registered. None of the recovering patients were vaccinated with any SARS-CoV-2 vaccine. Both clinics strictly required a negative PCR test for SARS-CoV-2 RNA detection 5 days before oocyte retrieval, except for those patients who were less than 3 months following recovery from SARS-Cov-2 infection. Patients in the control group were selected from medical records before March 2020 to ensure they did not have an infection and were not vaccinated.
Sampling Method: Non-Probability Sample
Enrollment: 428 (Actual)
Dates: Start 2021-12-12 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-09-18 (Actual)

PRIMARY OUTCOMES:
MII mature oocytes after retrieval | 2018 to 2022
Fertilization rate | 2018 to 2022
Blastocyst rate formation | 2018 to 2022

SECONDARY OUTCOMES:
antral follicular count before retrieval | 2018 to 2022

CONTACTS AND LOCATIONS:
Overall Officials: Jose A Moreno, PhD, Study Chair — Universitat Autonoma de Barcelona
Locations (1):
- Novafem, Bogotá, Colombia